CLINICAL TRIAL: NCT02864407
Title: A Regulatory Required Non Interventional Study to Monitor the Safety and Effectiveness of Once Daily Treatment of Orally Inhaled Vahelva Respimat (Tiotropium + Olodaterol Fixed Dose Combination 2.5µg/2.5µg Per Puff (2 Puffs Comprise One Medicinal Dose)) for Korean Patients With COPD (Chronic Obstructive Pulmonary Disease)
Brief Title: Vahelva Respimat Regulatory Post-marketing Surveillance in Korean Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237.60
Record Dates: First submitted 2016-07-20; First posted 2016-08-12 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vahelva® Respimat® (Tiotropium + Olodaterol fixed dose combination): Korean patients with COPD who are newly prescribed with Vahelva® Respimat® (Tiotropium + Olodaterol fixed dose combination).
  Interventions: Drug: Vahelva® Respimat® (Tiotropium + Olodaterol fixed dose combination)

INTERVENTIONS:
Drug: Vahelva® Respimat® (Tiotropium + Olodaterol fixed dose combination) — The recommended dose for adults is 5 microgram Tiotropium and 5 microgram Olodaterol given as two puffs from the Respimat® inhaler once daily at the same time of the day.

SUMMARY:
To monitor the safety profile and effectiveness of Vahelva Respimat in Korean patients with COPD in a routine clinical practice setting

DETAILED DESCRIPTION:
Study Design:

regulatory PMS study

ELIGIBILITY:
Inclusion criteria:

* Patients who have been started on Vahelva Respimat in accordance with the approved label in Korea
* Age >= 18 years at enrolment
* Patients who have signed on the data release consent form

Exclusion criteria:

* Patients with hypersensitivity to Vahelva Respimat or to any of the excipients.
* Patients with a history of hypersensitivity to atropine or its derivatives(e.g. ipratropium, oxitropium, glycopyrronium, clidinium, umeclidinium)
* Patients with asthma
* Current participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with COPD
Sampling Method: Probability Sample
Enrollment: 3223 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Chonnam National University Hospital, One Or Multiple Sites, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational prospective, non-interventional, open-label, multi-centre in Korean patients with Chronic Obstructive Pulmonary Disease (COPD).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination): Vahelva® Respimat® (Tiotropium + Olodaterol fixed dose combination) was prescribed according to the local label and at the discretion of the treating physician. The recommended dose for adults is 5 microgram Tiotropium and 5 microgram Olodaterol given as two puffs from the Respimat® inhaler once daily at the same time of the day. Each puff contains 2.5 microgram Tiotropium and 2.5 microgram Olodaterol.
Period: Overall Study
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Started (Enrolled) | 3223
Effectiveness Analysis Set | 2105
Long-term Safety Analysis Set | 813
Long-term Effectiveness Analysis Set | 767
Completed (Safety analysis set) | 3100
Not Completed | 123
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 115
Not completed — Not treated with Vahelva® Respimat® | 1
Not completed — Were administered Vahelva® Respimat® prior to the consent date | 3
Not completed — Consent prior to the contract date | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included those who signed the informed consent form to participate in this study as subject, took Vahelva® Respimat® once at least, and were completed follow up by the physician once or more.
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 3100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.14 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 425
  Male | 2675
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pre-dose percent predicted forced expiratory volume in one second (FEV1) [Mean (Standard Deviation); unit: percentage of predicted FEV1] — FEV1 is the maximum amount of air that can be forcefully exhaled in one second. It assesses the degree of airway obstruction in a routine test called spirometry, via a spirometer.
  FEVI was measured before the administration of Vahelva® Respimat® (pre-dose FEV1) at baseline. Pre-dose percent predicted FEV1 was calculated by converting the spirometer reading to a percentage of what would be predicted as normal FEV1 based on a several personal factors (e.g. sex, age, etc.). Population: Effectiveness Analysis Set included those who signed the informed consent form to participate in this study as subject, visited as per the study schedule, took Vahelva® Respimat® for 22 weeks ore more, the cases included in safety evaluation, and were evaluated for the effectiveness including overall evaluation (if the case assessed as 'unassessable' was excluded). Only participants with non-missing values are reported.
  percentage of predicted FEV1
    number analyzed (Participants) | 1127
    (all) | 58.38 (16.62)
Pre-dose percent predicted forced expiratory volume in one second (FEV1) [Mean (Standard Deviation); unit: percentage of predicted FEV1] — FEV1 is the maximum amount of air that can be forcefully exhaled in one second. It assesses the degree of airway obstruction in a routine test called spirometry, via a spirometer.
  FEVI was measured before the administration of Vahelva® Respimat® (pre-dose FEV1) at baseline. Pre-dose percent predicted FEV1 was calculated by converting the spirometer reading to a percentage of what would be predicted as normal FEV1 based on a several personal factors (e.g. sex, age, etc.). Population: Long-term effectiveness analysis set included those subjects in the safety analysis set who took Vahelva® Respimat® for 50 weeks or more. Only participants with non-missing values are reported.
  percentage of predicted FEV1
    number analyzed (Participants) | 418
    (all) | 57.75 (15.10)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Any Adverse Event, Unexpected Adverse Event, Unexpected Serious Adverse Event, Adverse Event Leading to Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An adverse event could therefore be any unfavourable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  An adverse event was assessed as unexpected if not listed in Local Product Information (LPI) and Company Core Data Sheet (CCDS).
  Percentage of subjects with any Adverse Event, unexpected Adverse Event, unexpected Serious Adverse Event, Adverse Event leading to discontinuation is reported. Percentages were rounded to two decimal places.
Time Frame: From the signing date on Informed Consent Form (ICF) to 28 days after last administration date of Vahelva® Respimat®, up to 52 (±2) weeks+ 28 days.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 3100
percentage of participants
  Any Adverse Event | 19.90 [18.51 to 21.35]
  Unexpected Adverse Event | 13.65 [12.46 to 14.90]
  Unexpected Serious Adverse Event | 3.48 [2.87 to 4.19]
  Adverse Event leading to discontinuation | 2.29 [1.79 to 2.88]

2. Primary Outcome: Percentage of Subjects With Any Adverse Drug Reaction, Serious Adverse Drug Reaction, Unexpected Adverse Drug Reaction, Unexpected Serious Adverse Drug Reaction, Adverse Drug Reaction Leading to Discontinuation
Description: An adverse drug reaction (ADR) was defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility. Adverse reactions may arise from use of the product within or outside the terms of the marketing authorization or from occupational exposure. Conditions of use outside the marketing authorization include off label use, overdose, misuse, abuse and medication errors. Investigator was primarily responsible to assess ADR relatedness.
  An ADR was assessed as unexpected if not listed in Local Product Information (LPI) and Company Core Data Sheet (CCDS).
  Percentage of subjects with any Adverse Drug Reaction, serious Adverse Drug Reaction, unexpected Adverse Drug Reaction, unexpected Serious Adverse Drug Reaction, Adverse Drug Reaction leading to discontinuation is reported. Percentages were rounded to two decimal places.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 3100
percentage of participants
  Any Adverse Drug Reaction | 2.87 [2.31 to 3.52]
  Serious Adverse Drug Reaction | 0.16 [0.05 to 0.38]
  Unexpected Adverse Drug Reaction | 1.16 [0.81 to 1.60]
  Unexpected Serious Adverse Drug Reaction | 0.13 [0.04 to 0.33]
  Adverse Drug Reaction leading to discontinuation | 1.32 [0.95 to 1.79]

3. Primary Outcome: Percentage of Subjects With Any Adverse Event (AE) in the Long-term Safety Analysis Set
Description: An adverse event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An adverse event could therefore be any unfavourable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  Percentage of participants with any AE is reported. Percentages were rounded to two decimal places.
Time Frame: as for outcome 1
Population: Long term safety analysis set included those subjects in the safety analysis set who took Vahelva® Respimat® for 50 weeks or more.
Measure: Number (95% Confidence Interval); unit: percentage of partcipants
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 813
percentage of partcipants | 22.88 [20.03 to 25.92]

4. Primary Outcome: Change From Baseline in Pre-dose Percent Predicted Forced Expiratory Volume in One Second (FEV1) to Week 24 in the Effectiveness Analysis Set
Description: FEV1 is the maximum amount of air that can be forcefully exhaled in one second. It assesses the degree of airway obstruction in a routine test called spirometry, via a spirometer. FEVI was measured before the administration of Vahelva® Respimat® (pre-dose FEV1) at baseline and at Week 24 (±2 weeks). Pre-dose percent predicted FEV1 was calculated by converting the spirometer reading to a percentage of what would be predicted as normal FEV1 based on a several personal factors (e.g. sex, age, etc.).
  Change from baseline in pre-dose percent predicted FEV1 to Week 24 was calculated as: pre-dose percent predicted FEV1 value at Week 24 (±2 weeks) - pre-dose percent predicted FEV1 value at baseline.
Time Frame: At baseline (30 days before baseline visit (Visit 1)) and Week 24 (±2 weeks).
Population: Effectiveness analysis set included those who signed the informed consent form to participate in this study as subject, visited as per the study schedule, took Vahelva® Respimat® for 22 weeks or more, the cases included in safety evaluation, and were evaluated for the effectiveness including overall evaluation (if the case assessed as 'unassessable' was excluded). Only participants with non-missing values are reported.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 450
percentage of predicted FEV1 | 5.41 (9.63)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test — p-value for difference of Follow-up Week 24 (±2weeks) versus Baseline

5. Primary Outcome: Change From Baseline in Pre-dose Percent Predicted Forced Expiratory Volume in One Second (FEV1) to Week 52 in the Effectiveness Analysis Set
Description: FEV1 is the maximum amount of air that can be forcefully exhaled in one second. It assesses the degree of airway obstruction in a routine test called spirometry, via a spirometer. FEVI was measured before the administration of Vahelva® Respimat® (pre-dose FEV1) at baseline and at Week 52 (±2 weeks). Pre-dose percent predicted FEV1 was calculated by converting the spirometer reading to a percentage of what would be predicted as normal FEV1 based on a several personal factors (e.g. sex, age, etc.).
  Change from baseline in pre-dose percent predicted Forced Expiratory Volume in one second (FEV1) to Week 52 was calculated as: pre-dose percent predicted FEV1 value at Week 52 (±2 weeks) - pre-dose percent predicted FEV1 value at baseline.
Time Frame: At baseline (30 days before baseline visit (Visit 1)) and Week 52 (±2 weeks).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 231
percentage of predicted FEV1 | 4.91 (10.00)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test — p-value for difference of Week 52 (±2 weeks) versus Baseline

6. Primary Outcome: Change From Baseline in Pre-dose Percent Predicted Forced Expiratory Volume in One Second (FEV1) to Week 24 in the Long-term Effectiveness Analysis Set
Description: FEV1 is the maximum amount of air that can be forcefully exhaled in one second. It assesses the degree of airway obstruction in a routine test called spirometry, via a spirometer. FEVI was measured before the administration of Vahelva® Respimat® (pre-dose FEV1) at baseline and at Week 24 (±2 weeks). Pre-dose percent predicted FEV1 was calculated by converting the spirometer reading to a percentage of what would be predicted as normal FEV1 based on a several personal factors (e.g. sex, age, etc.).
  Change from baseline in pre-dose percent predicted Forced Expiratory Volume in one second (FEV1) to Week 24 was calculated as: pre-dose percent predicted FEV1 value at Week 24 (±2 weeks) - pre-dose percent predicted FEV1 value at baseline.
Time Frame: At baseline (30 days before baseline visit (Visit 1)) and Week 24 (±2 weeks).
Population: Long-term effectiveness analysis set included those subjects in the safety analysis set who took Vahelva® Respimat® for 50 weeks or more. Only participants with non-missing values are reported.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 169
percentage of predicted FEV1 | 6.13 (9.29)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test — p-value for difference of Follow-up Week 24 (±2weeks) versus Baseline

7. Primary Outcome: Change From Baseline in Pre-dose Percent Predicted Forced Expiratory Volume in One Second (FEV1) to Week 52 in the Long-term Effectiveness Analysis Set
Description: as for outcome 5
Time Frame: At baseline (30 days before baseline visit (Visit 1)) and Week 52 (±2 weeks).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 195
percentage of predicted FEV1 | 4.83 (10.34)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test — p-value for difference of Follow-up Week 52 (±2weeks) versus Baseline

8. Secondary Outcome: Change From Baseline in Post Bronchodilator Percent Predicted Forced Expiratory Volume in One Second (FEV1) to Week 24 in the Effectiveness Analysis Set
Description: FEV1 is the maximum amount of air that can be forcefully exhaled in one second. FEVI was measured via a spirometer after the administration of the bronchodilator (Vahelva® Respimat®) at baseline and at Week 24 (±2 weeks). Post bronchodilator percent predicted FEV1 was calculated by converting the spirometer reading to a percentage of what would be predicted as normal FEV1 based on a several personal factors (e.g. sex, age, etc.).
  Change from baseline in post bronchodilator percent predicted FEV1 to Week 24 was calculated as: post bronchodilator percent predicted FEV1 value at Week 24 (±2 weeks) - post bronchodilator percent predicted FEV1 value at baseline.
Time Frame: At baseline and Week 24 (±2 weeks).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 480
percentage of predicted FEV1 | 3.80 (8.83)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test; p-value for difference of Follow-up Week 24 (±2weeks) versus Baseline

9. Secondary Outcome: Change From Baseline in Post Bronchodilator Percent Predicted Forced Expiratory Volume in One Second (FEV1) to Week 52 in the Effectiveness Analysis Set
Description: FEV1 is the maximum amount of air that can be forcefully exhaled in one second. FEVI was measured via a spirometer after the administration of the bronchodilator (Vahelva® Respimat®) at baseline and at Week 52 (±2 weeks). Post bronchodilator percent predicted FEV1 was calculated by converting the spirometer reading to a percentage of what would be predicted as normal FEV1 based on a several personal factors (e.g. sex, age, etc.).
  Change from baseline in post bronchodilator percent predicted FEV1 to Week 52 was calculated as: post bronchodilator percent predicted FEV1 value at Week 52 (±2 weeks) - post bronchodilator percent predicted FEV1 value at baseline.
Time Frame: At baseline and Week 52 (±2 weeks).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 230
percentage of predicted FEV1 | 4.52 (9.23)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test; p-value for difference of Follow-up Week 52 (±2weeks) versus Baseline

10. Secondary Outcome: Change From Baseline in Post Bronchodilator Percent Predicted Forced Expiratory Volume in One Second (FEV1) to Week 24 in the Long-term Effectiveness Analysis Set
Description: as for outcome 8
Time Frame: At baseline and Week 24 (±2 weeks).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 135
percentage of predicted FEV1 | 5.19 (8.80)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test; p-value for difference of Follow-up Week 24 (±2weeks) versus Baseline

11. Secondary Outcome: Change From Baseline in Post Bronchodilator Percent Predicted Forced Expiratory Volume in One Second (FEV1) to Week 52 in the Long-term Effectiveness Analysis Set
Description: as for outcome 9
Time Frame: At baseline and Week 52 (±2 weeks).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 200
percentage of predicted FEV1 | 4.36 (9.16)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test; p-value for difference of Follow-up Week 52 (±2weeks) versus Baseline

12. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score at Week 24 in the Effectiveness Analysis Set
Description: Transition dyspnea index (TDI) is a validated, interviewer-administered questionnaire that measures changes in dyspnea severity from the baseline. TDI consists of 3 individual components: functional impairment, magnitude of task, and magnitude of effort. Each component was rated by 7 grades from -3 (major deterioration) to +3 (major improvement), and were sum up to form a TDI focal score from -9 to +9, with higher scores indicating better outcomes.
Time Frame: At Week 24 (±2 weeks).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 585
units on a scale | -0.18 (0.64)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test — p-value for difference of Week 24 (±2 weeks) versus Baseline

13. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score at Week 52 in the Effectiveness Analysis Set
Description: as for outcome 12
Time Frame: At Week 52 (±2 weeks).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 137
units on a scale | -0.39 (0.79)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test — p-value for difference of 52±2 weeks versus Baseline

14. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score at Week 24 in the Long-term Effectiveness Analysis Set
Description: as for outcome 12
Time Frame: At Week 24 (±2 weeks).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 134
units on a scale | -0.31 (0.63)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test — p-value for difference of Week 24 (±2 weeks) versus Baseline

15. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score at Week 52 in the Long-term Effectiveness Analysis Set
Description: as for outcome 12
Time Frame: At Week 52 (±2 weeks).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 110
units on a scale | -0.44 (0.78)
Statistical Analysis 1: Comparison: Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination); Test type: Other; p < 0.0001, Paired t-test — p-value for difference of Week 52 (±2 weeks) versus Baseline

16. Secondary Outcome: Number of Subjects in Each Category of Overall Evaluation in the Effectiveness Analysis Set
Description: Overall evaluation (improved, unchanged or aggravated) was performed by investigator and was based on overall clinical assessment including change from baseline in effectiveness assessment (pre-dose percent predicted Forced Expiratory Volume in one second (FEV1), post bronchodilator percent predicted Forced Expiratory Volume in one second (FEV1), Transition dyspnea index (TDI)) after 24 weeks or 52 weeks of treatment.
  Improved, unchanged, aggravated are defined as below:
  * Improved : If determined as there is any effect of maintaining or improving symptoms;
  * Unchanged : If symptoms have not been changed compared with before and not determined as there is any effect of maintaining symptoms;
  * Aggravated : If symptoms are worse than before administration. Number of subject in each category of overall evaluation (improved, unchanged or aggravated) is reported.
Time Frame: At baseline and at Week 24 (±2 weeks) or at Week 52 (±2 weeks).
Population: Effectiveness analysis set included those who signed the informed consent form to participate in this study as subject, visited as per the study schedule, took Vahelva® Respimat® for 22 weeks or more, the cases included in safety evaluation, and were evaluated for the effectiveness including overall evaluation (if the case assessed as 'unassessable' was excluded).
Measure: Count of Participants; unit: Participants
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 2105
Participants
  Improved | 1386
  Unchanged | 711
  Aggravated | 8

17. Secondary Outcome: Number of Subjects in Each Category of Overall Evaluation in the Long-term Effectiveness Analysis Set
Description: as for outcome 16
Time Frame: At baseline and at Week 24 (±2 weeks) or at Week 52 (±2 weeks).
Population: Long-term effectiveness analysis set included those subjects in the safety analysis set who took Vahelva® Respimat® for 50 weeks or more.
Measure: Count of Participants; unit: Participants
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 767
Participants
  Improved | 543
  Unchanged | 220
  Aggravated | 4
  Unassessable | 0

18. Secondary Outcome: Effectiveness Rate in the Effectiveness Analysis Set
Description: Overall evaluation (Improved, unchanged or aggravated) by investigator was based on overall clinical assessment including change from baseline in effectiveness assessment (pre-dose percent predicted Forced Expiratory Volume in one second (FEV1), post bronchodilator percent predicted Forced Expiratory Volume in one second (FEV1), Transition dyspnea index (TDI)) after 24 weeks or 52 weeks of treatment. 'Improved' was assessed as "Effective", 'Unchanged, Aggravated' were assessed as "Invalid".
Time Frame: At baseline and at Week 24 (±2 weeks) or at Week 52 (±2 weeks).
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 2105
percentage of participants | 65.84 [63.77 to 67.87]

19. Secondary Outcome: Effectiveness Rate in the Long-term Effectiveness Analysis Set
Description: Overall evaluation (Improved, unchanged, aggravated or unassessable) by investigator was based on overall clinical assessment including change from baseline in effectiveness assessment (pre-dose percent predicted Forced Expiratory Volume in one second (FEV1), post bronchodilator percent predicted Forced Expiratory Volume in one second (FEV1), Transition dyspnea index (TDI)) after 24 weeks or 52 weeks of treatment. 'Improved' was assessed as "Effective", 'Unchanged, Aggravated' were assessed as "Invalid".
Time Frame: At baseline and at Week 24 (±2 weeks) or at Week 52 (±2 weeks).
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
Number analyzed (Participants) | 767
percentage of participants | 70.80 [67.44 to 73.99]

ADVERSE EVENTS:
Time Frame: From the signing date on Informed Consent Form (ICF) to 28 days after last administration date of medication, up to 52 (±2) weeks+ 28 days.
Description: Safety Analysis Set included those who signed the informed consent form to participate in this study as subject, took Vahelva® Respimat® once at least, and were completed follow up by the physician once or more.
Arm/Group | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination)
All-Cause Mortality (participants affected / at risk) | 12/3100
Serious Adverse Events (participants affected / at risk) | 147/3100
Other Adverse Events (participants affected / at risk) | 0/3100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vahelva® Respimat® (Tiotropium + Olodaterol Fixed Dose Combination) (N=3100)
Coagulopathy (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Arteriospasm coronary (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cor pulmonale (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Cataract (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 1
Post procedural complication (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Death (General disorders) | 1
Pyrexia (General disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Bronchiolitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Mycobacterial infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 30
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia influenzal (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bell's palsy (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 4
Metabolic encephalopathy (Nervous system disorders) | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02864407/Prot_SAP_000.pdf